CLINICAL TRIAL: NCT03029806
Title: Lysine-specific Demethylase 1 and Salt-sensitivity in Humans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan S. Williams, MD, MMSc, Associate Physician, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015P002540
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Vascular Stiffness

STUDY DESIGN:
Intervention Model Description: Heathy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Afr-Amer risk allele (Active Comparator): African Americans carrying the LSD1 affected allele
  Interventions: Other: Aldosterone response to AngII LS; Other: Renal blood flow response to salt; Other: Vascular Stiffness
- Cauc risk allele (Placebo Comparator): Caucasians carrying the LSD1 affected allele
  Interventions: Other: Aldosterone response to AngII LS; Other: Renal blood flow response to salt; Other: Vascular Stiffness
- Afr-Amer non-risk allele (Placebo Comparator): African Americans carrying the LSD1 non-risk allele
  Interventions: Other: Aldosterone response to AngII LS; Other: Renal blood flow response to salt; Other: Vascular Stiffness
- Cauc non-risk allele (Placebo Comparator): Caucasians carrying the LSD1 non-risk allele
  Interventions: Other: Aldosterone response to AngII LS; Other: Renal blood flow response to salt; Other: Vascular Stiffness

INTERVENTIONS:
Other: Aldosterone response to AngII LS — Change in aldosterone from baseline to after Ang II infusion on a LS diet
Other: Renal blood flow response to salt — Change in renal blood flow: High salt to low salt diet
Other: Vascular Stiffness — Change in vascular stiffness, baseline compared to AngII

SUMMARY:
The purpose of this study is to investigate the role dietary salt plays in epigenetic regulation of blood pressure, focusing on the salt-sensitive regulatory enzyme Lysine-specific demethylase 1.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role dietary salt plays in epigenetic regulation of blood pressure in African American and Caucasians, focusing on the salt-sensitive regulatory enzyme Lysine-specific demethylase 1. This might help us understand why some people develop high blood pressure.

Healthy volunteers will be screened for eligibility and invited to participate in a 2 weeks study. Week 1 will be consumption of a low salt diet. Week 2 will be a high salt diet.

At the end of each week, participants will be admitted to a Clinical Research Center overnight and for one day.

On the CRC, participants will remain fasting and supine overnight and then next morning undergo hormonal and vascular testing. This will consist of blood drawing, echocardiogram, vascular tonometry, and assessment of renal blood flow before and after a low-dose Angiotensin II infusion.

The study outcome will compare how variants in the LSD1 gene affect hormonal and vascular responses according to race. This information will help us determine why some races and genetic profiles are more susceptible to detrimental effects of salt in the diet while others are protected against these effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-45 years
* Caucasian or African American
* No gender preference (anticipate 50% female)
* Normotensive (screening blood pressure <140/90 mmHg)
* No history of hypertension, diabetes, stroke, coronary artery disease, kidney disease, cancer, thyroid disease, preeclampsia, or hospitalizations in 6 months
* Normal screening laboratory values (CMP, TSH, A1c)
* Normal ECG
* BMI <25 kg/m2

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Any medication or herbal preparation
* >6oz alcohol/week
* Tobacco use
* Illicit drug use
* Chronic NSAID use
* Recent steroid use (injected, inhaled, oral)
* Decongestant use in the past 2 weeks
* Known sensitivity to infused Angiotensin II or para-amino hippurate

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Aldosterone response to angiotensin II | After 1 week dietary salt manipulation
  Change in aldosterone, baseline to after angiotensin II by genotype/race

SECONDARY OUTCOMES:
Renal blood flow response to dietary salt | After 1 week dietary salt manipulation on both diets
  Change in renal blood flow, high salt diet to low salt diet by genotype/race
Vascular stiffness response to angiotensin II | After 1 week dietary salt manipulation
  Change in vascular stiffness, baseline to after angiotensin II by genotype/race

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared first thru the publication of research results in peer-review scientific journals by the study investigator. IPD will be made available upon reasonable request from bona fide research organizations in an effort to provide broader impact and enrich public health knowledge. Research volunteer PHI will not be shared, and all participant data will be de-identified and coded. Only encrypted and secure network exchanges will be used for data transfer. Cost sharing my be required in order prepare datasets.

REFERENCES:
- [Background] Krug AW, Tille E, Sun B, Pojoga L, Williams J, Chamarthi B, Lichtman AH, Hopkins PN, Adler GK, Williams GH. Lysine-specific demethylase-1 modifies the age effect on blood pressure sensitivity to dietary salt intake. Age (Dordr). 2013 Oct;35(5):1809-20. doi: 10.1007/s11357-012-9480-0. Epub 2012 Oct 2. PMID 23054827
- [Background] Williams JS, Chamarthi B, Goodarzi MO, Pojoga LH, Sun B, Garza AE, Raby BA, Adler GK, Hopkins PN, Brown NJ, Jeunemaitre X, Ferri C, Fang R, Leonor T, Cui J, Guo X, Taylor KD, Ida Chen YD, Xiang A, Raffel LJ, Buchanan TA, Rotter JI, Williams GH, Shi Y. Lysine-specific demethylase 1: an epigenetic regulator of salt-sensitive hypertension. Am J Hypertens. 2012 Jul;25(7):812-7. doi: 10.1038/ajh.2012.43. Epub 2012 Apr 26. PMID 22534796
- [Background] Pojoga LH, Williams JS, Yao TM, Kumar A, Raffetto JD, do Nascimento GR, Reslan OM, Adler GK, Williams GH, Shi Y, Khalil RA. Histone demethylase LSD1 deficiency during high-salt diet is associated with enhanced vascular contraction, altered NO-cGMP relaxation pathway, and hypertension. Am J Physiol Heart Circ Physiol. 2011 Nov;301(5):H1862-71. doi: 10.1152/ajpheart.00513.2011. Epub 2011 Aug 26. PMID 21873498
- [Derived] Heydarpour M, Parksook WW, Pojoga LH, Williams GH, Williams JS. Mineralocorticoid Receptor and Aldosterone: Interaction Between NR3C2 Genetic Variants, Sex, and Age in a Mixed Cohort. J Clin Endocrinol Metab. 2024 Dec 18;110(1):e140-e149. doi: 10.1210/clinem/dgae127. PMID 38437868